CLINICAL TRIAL: NCT05459298
Title: Randomized Trial of Enteral Vitamin D Supplementation in Infants < 28 Weeks Gestational Age or <1000 Grams Birth Weight
Brief Title: ViDES Trial (Vitamin D Extra Supplementation)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Maria del Mar Romero López, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HSC-MS-22-0563; KL2TR003168 (NIH); R03TR005545 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Vitamin D Deficiency
Keywords: Premature infant; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Premature Birth | interventions — Saline Solution; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus placebo (Active Comparator): Infants will receive placebo (normal saline) in the first 28 days after birth. Care will be unaffected and provided based on the judgment of the attending neonatal faculty and NICU policies and routine practices. When the infant receives about 120 to 160 mL/kg/day of fortified milk at 24 kcal/ounce, the infant will receive supplementation with 400 IU/day of vitamin D as usual care.
  Interventions: Dietary Supplement: Placebo; Other: Usual Care
- Usual care plus vitamin D supplementation (Experimental): Infants will receive cholecalciferol 800 IU/day in the first 28 days after birth, given enterally four times per day (0.5mL per dose = 200 IU) until the infant is provided 400 IU/day (when feedings reach about 120 -160 mL/kg/day). At that point the study cholecalciferol will be reduced to 400 IU/day for a total supplementation of 800 IU/day.
  Interventions: Dietary Supplement: 800 IU/day vitamin D supplementation with feedings in the first 28 days after birth; Other: Usual Care

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo is normal saline, given in the first 28 days after birth, prepared to have the same volume and appearance as vitamin D, which is a clear odorless solution.
  Other Names: Normal saline
  Arms: Usual care plus placebo
Dietary Supplement: 800 IU/day vitamin D supplementation with feedings in the first 28 days after birth — 800 IU/day Vitamin D supplementation until 400 IU/day are provided as part of usual care (started when infants receive full feedings of about 120-160 mL/kg/day). At that point the intervention becomes a supplement of 400 IU/day above that given with usual care. In this way all infants in the intervention group receive 800 IU/day of vitamin D total supplementation in the first 28 days after birth with feedings.
  Other Names: Cholecalciferol
  Arms: Usual care plus vitamin D supplementation
Other: Usual Care — Care will be unaffected and provided based on the judgment of the attending neonatal faculty and NICU policies and routine practices. When the infant receives about 120 to 160 mL/kg/day of fortified milk at 24 kcal/ounce, the infant will receive supplementation with 400 IU/day of vitamin D as usual care.

SUMMARY:
The objective of the study is to compare supplementation with vitamin D at 800 IU/day to usual care for the first 28 days after birth with respect to 25 (OH) vitamin D levels and indicators of likely or plausible effects of vitamin D supplementation on the function or structure of the lung, bones, immune system, and brain in extremely premature (EP) infants who are <28 weeks gestational age (GA) or <1000 grams of birth weight (BW). The study results will be analyzed as intention to treat Bayesian analyses (Frequentist analyses will also be performed).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at < 28 weeks gestational age (GA) or <1000 grams birth weight (BW)
* Inborn
* Informed written consent in an Institutional Review Board (IRB)-approved manner

Exclusion Criteria:

* GA >32 weeks regardless of birth weight (BW)
* Any major congenital anomaly
* A known congenital nonbacterial infection
* Prenatal diagnosis of disorders that affect vitamin D absorption (e.g, cystic fibrosis)
* Such severe illness or immaturity that the attending neonatologist judges intensive care to be unjustified.

Ages: 24 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
25-hydroxyvitamin D (25[OH]D) level | about 28 days after birth

SECONDARY OUTCOMES:
25-hydroxyvitamin D (25[OH]D) level | 36 weeks after birth
Type of respiratory support required at 36 weeks postmenstrual age | 36 weeks postmenstrual age (or at the time of discharge home if earlier)
  Data will be reported categorically as:
  * Number of participants who survive without respiratory support
  * Number of participants who survive with nasal cannula at ≤ 2 liters (L)/minute
  * Number of participants who survive with nasal cannula >2 L/minute or noninvasive positive airway pressure
  * Number of participants who survive with invasive mechanical ventilation
  * Number of participants who die
Length of Hospital stay | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of participants who are still on respiratory support | 22 to 26 months corrected age
  Respiratory support includes supplemental oxygen and positive pressure ventilation.
Number of days of supplemental oxygen | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of days of mechanical ventilation | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of days of positive pressure support | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of participants who receive steroid treatment to decrease respiratory support | from baseline to 36 weeks postmenstrual age
Number of participants with pulmonary hypertension | 36 weeks postmenstrual age
Number of participants with recurrent wheezing | 2 years
  Assessed using the validated International Study of Asthma and Allergies modified asthma scale, which is defined as having more than two episodes (with or without a documented respiratory tract infection) in the 6 months before the 2-year-old visit
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Number of participants with any fractures | from baseline to 36 weeks postmenstrual age
Number of participants with hospital-acquired sepsis | from day 3 after birth to the time of discharge (which is 0 to 60 weeks after birth)
Calcium level | 0 to 36 weeks postmenstrual age
Phosphorus level | 0 to 36 weeks postmenstrual age
Alkaline phosphatase level | 0 to 36 weeks postmenstrual age
Neurodevelopment as assessed by the Bayley-IV Scales of Infant and Toddler Development | 2 years
  Score ranges from 40 to 160, with a higher score indicating a better outcome.
Number of participants with neurodevelopmental impairment (NDI) | 2 years
Number of participants who die or have a morbidity | 36 weeks postmenstrual age
  Morbidities include retinopathy of prematurity (ROP), intraventricular hemorrhage (IVH), bronchopulmonary dysplasia (BPD), neurodevelopmental impairment (NDI), necrotizing enterocolitis (NEC), and patent ductus arteriosus (PDA).
Vitamin D status as indicated by serum concentration of 24,25(OH)2D3 as assessed by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) | about 28 days after birth
Vitamin D status as indicated by serum concentration of 24,25(OH)2D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age
Vitamin D status as indicated by serum concentration of 3-epi-25(OH)D3 as assessed by LC-MS/MS | about 28 days after birth
Vitamin D status as indicated by serum concentration of 3-epi-25(OH)D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age
Vitamin D status as indicated by serum concentration of 25(OH)D3 as assessed by LC-MS/MS | about 28 days after birth
Vitamin D status as indicated by serum concentration of 25(OH)D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age
Pre-discharge health system costs | From time of birth to time of discharge (about 0 to 60 weeks after birth)
  Facility costs will be extracted from the hospital's cost-accounting systems. Costs associated with physician services during the birth admission will be estimated using CPT-based claims data and Relative Value Units (RVUs) from the Medicare Fee Schedule. The cost of oral vitamin D will be determined using the average wholesale price listed in the Micromedex RedBook
Cost-effectiveness in preventing days of respiratory support | From time of birth to time of discharge (about 0 to 60 weeks after birth)
  Incremental health system costs per prevented day of respiratory support
Cost-effectiveness in increasing survival without BPD | From time of birth to time of discharge (about 0 to 60 weeks after birth)
  Incremental health system costs per prevented day of respiratory support

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Mar Romero López, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romero-Lopez M, Tyson JE, Naik M, Pedroza C, Holzapfel LF, Avritscher E, Mosquera R, Khan A, Rysavy M. Randomized Controlled Trial of Enteral Vitamin D Supplementation (ViDES) in Infants <28 Weeks Gestational Age or <1000 Grams Birth Weight: Study Protocol. Res Sq [Preprint]. 2024 Jun 25:rs.3.rs-4049246. doi: 10.21203/rs.3.rs-4049246/v1. PMID 38978597
- [Derived] Romero-Lopez M, Tyson JE, Naik M, Pedroza C, Holzapfel LF, Avritscher E, Mosquera R, Khan A, Rysavy M. Randomized controlled trial of enteral vitamin D supplementation (ViDES) in infants <28 weeks gestational age or <1000 g birth weight: study protocol. Trials. 2024 Jun 28;25(1):423. doi: 10.1186/s13063-024-08274-8. PMID 38943179